CLINICAL TRIAL: NCT05073406
Title: Cognitive Performance After Acute Exposure to Altitude - Part II
Brief Title: Cognition at Altitude in HEMS - Part II
Acronym: HEMS II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mountain Emergency Medicine (Other)
Collaborators: University Grenoble Alps (Other); Università degli Studi di Trento (Other); Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Giacomo Strapazzon, MD PhD, Principal Investigator, Institute of Mountain Emergency Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 98-2021
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-01

CONDITIONS: Hypobaric Hypoxia; Hypobaric Normoxia; Cognitive Performance; Emergency Medicine; Stress Physiology

STUDY DESIGN:
Intervention Model Description: Interventional, non-pharmacological, randomized, controlled, double-blinded, cross-over
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypobaric normoxia (Experimental): Altitude exposure in hypobaric normoxic condition
  Interventions: Other: Altitude exposure in hypobaric normoxic condition
- Hypobaric hypoxia (Sham Comparator): Altitude exposure in hypobaric hypoxic condition
  Interventions: Other: Altitude exposure in hypobaric hypoxic condition

INTERVENTIONS:
Other: Altitude exposure in hypobaric normoxic condition — Altitude exposure with oxygen supplementation to achieve normoxia at altitude
  Arms: Hypobaric normoxia
Other: Altitude exposure in hypobaric hypoxic condition — Altitude exposure with air supplementation to obtain a sham comparator arm
  Arms: Hypobaric hypoxia

SUMMARY:
The aim of the current study is to evaluate under blinded conditions, both in a simulated environment and during helicopter flight, the effect of a rapid (within 20 minutes) exposure to altitude (4000 m asl) on physiological parameters and selected cognitive domains, in providers operating in helicopter emergency medical service (HEMS) exposed to hypobaric hypoxia or to hypobaric normoxia (H0: cognitive effects under hypobaric hypoxia = cognitive effects under hypobaric normoxia). Simulated environment will allow to control different factors. The parallelism between a study branch conducted in a simulated environment and another one conducted under a real-life condition will allow to evaluate the additive effects on additional stressor factors (processive and systemic ones).

* Simulation branch: each participant will take part in three research sessions: a familiarization session and two experimental sessions in simulation facility called terraXcube (test 1 and 2). On test 1 and test 2 each group will be exposed twice to the simulated altitude of 4000 m asl (under hypobaric hypoxia or hypobaric normoxia conditions) according to the randomization protocol. Participants will perform the neurocognitive tests three times on each of the two tests: before the ascent (TC0), after 5 min from the end of the ascent (TC1) and after around 30 min (TC2), to investigate European Union Aviation Safe Agency (EASA) proposed recommendations. After completing each neurocognitive test session, participants will be asked to rate their performance using a visual analogue scales (VAS). All participants will wear the vital parameters monitoring system during the entire duration of the tests inside the chamber, as well as the cerebral oxygen saturation (ScO2) sensor. Samples will be collected by saliva, urine and/or capillary blood. The same schedule is repeated in each test session.
* In-field branch: each participant will take part in three research sessions: a familiarization session and two experimental sessions during helicopter flights (test 1 and 2). On test 1 and test 2 each group will be exposed twice to the altitude of 4000 m (under hypobaric hypoxia or hypobaric normoxia conditions) according to the randomization protocol. Participants will perform the neurocognitive test two times on each test: before the ascent (TC0), after around 5 min from the end of the ascent (TC1). After completing each neurocognitive tests, participants will be asked to rate their performance using a visual analogue scales (VAS). All participants will wear the vital parameters monitoring system during the entire duration of the tests. Samples will be collected. The same schedule is planned in each test session.

ELIGIBILITY:
Inclusion Criteria:

* members of emergency medical services (EMS) and search and rescue (SAR) services with an occupational licence;
* an age between 18 and 60 years;
* an American Society of Anaesthesiologists (ASA) physical status class I;
* provided informed and written consent;
* no current COVID 19 symptoms and temperature ≤ 37.5°on test days, not being tested positive for COVID-19, ideally COVID-19 vaccinated.

Exclusion Criteria:

* members under the age of 18 years;
* an ASA physical status class II or more;
* a medical history of psychiatric disorders and neurological diseases;
* previous high altitude pulmonary oedema (HAPE) or high altitude cerebral oedema (HACE) or severe acute mountain sickness (AMS) (defined as a Lake Louise Score (LLS) > 9) occurred at altitudes similar to the ones tested in the study;
* no informed consent;
* current COVID 19 symptoms, being tested positive for COVID-19 or symptoms and body temperature ≥ 37.5°on test days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Psychomotor Vigilance Test - PVT | Changes from baseline (T0) to altitude measurement (respectively after 5 min - T1 and after 30 min - T2)
  Changes in reaction time using a computer-based test (PVT)
Digit-Symbol Substitution Task - DSST | Changes from baseline (TC0) to altitude measurement (respectively after 5 min - TC1 and after 30 min - TC2)
  Changing in processing speed using a computer based test (DSST)
2-back Test | Changes from baseline (TC0) to altitude measurement (respectively after 5 min - TC1 and after 30 min - TC2)
  Changing in working memory using a computer based test (2-back test)

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Strapazzon, MD PhD, Principal Investigator — Eurac Research, Institute of Mountain Emergency Medicine; Marika Falla, MD PhD, Principal Investigator — University of Trento, Center for Mind/Brain Sciences - CIMeC; Michiel van Veelen, MD, Principal Investigator — Eurac Research, Institute of Mountain Emergency Medicine
Locations (1):
- Eurac Research, Institute of Mountain Emergency Medicine, Bolzano, BZ, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Basner M, Moore TM, Nasrini J, Gur RC, Dinges DF. Standardization of psychomotor vigilance testing methods and reporting. Sleep. 2021 Jul 9;44(7):zsab114. doi: 10.1093/sleep/zsab114. No abstract available. PMID 34019081
- [Background] Brodmann Maeder M, Brugger H, Pun M, Strapazzon G, Dal Cappello T, Maggiorini M, Hackett P, Bartsch P, Swenson ER, Zafren K. The STAR Data Reporting Guidelines for Clinical High Altitude Research. High Alt Med Biol. 2018 Mar;19(1):7-14. doi: 10.1089/ham.2017.0160. Epub 2018 Feb 9. PMID 29596018
- [Background] Cable GG. In-flight hypoxia incidents in military aircraft: causes and implications for training. Aviat Space Environ Med. 2003 Feb;74(2):169-72. PMID 12602449
- [Background] EASA. https://www.easa.europa.eu/document-library/notices-of-proposed-amendment/npa-2018-04. (2018).
- [Background] Falla M, Papagno C, Dal Cappello T, Vogele A, Hufner K, Kim J, Weiss EM, Weber B, Palma M, Mrakic-Sposta S, Brugger H, Strapazzon G. A Prospective Evaluation of the Acute Effects of High Altitude on Cognitive and Physiological Functions in Lowlanders. Front Physiol. 2021 Apr 28;12:670278. doi: 10.3389/fphys.2021.670278. eCollection 2021. PMID 33995130
- [Background] Falla M, Hufner K, Falk M, Weiss EM, Vogele A, Jan van Veelen M, Weber B, Brandner J, Palma M, Dejaco A, Brugger H, Strapazzon G. Simulated Acute Hypobaric Hypoxia Effects on Cognition in Helicopter Emergency Medical Service Personnel - A Randomized, Controlled, Single-Blind, Crossover Trial. Hum Factors. 2024 Feb;66(2):404-423. doi: 10.1177/00187208221086407. Epub 2022 May 31. PMID 35640630
- [Background] Hart, S., and Staveland, L. (1988). "Development of NASA-TLX (task load index) - results ofempirical and theoretical research," in HumanMental Workload, eds P. Hancock and N. Meshkati (Amsterdam: Springer), 139-183. doi: 10.1016/ s0166- 4115(08)62386- 9.
- [Background] Hinkelbein J, Glaser E. Evaluation of two oxygen face masks with special regard to inspiratory oxygen fraction (FiO2) for emergency use in rescue helicopters. Air Med J. 2008 Mar-Apr;27(2):86-90. doi: 10.1016/j.amj.2007.07.005. PMID 18328973
- [Background] Mrakic-Sposta S, Vezzoli A, Malacrida S, Falla M, Strapazzon G. "Direct" and "Indirect" Methods to Detect Oxidative Stress During Acute or Chronic High-Altitude Exposure. High Alt Med Biol. 2017 Sep;18(3):303-304. doi: 10.1089/ham.2017.0067. Epub 2017 Jul 28. No abstract available. PMID 28753037
- [Background] Nowacki J, Heekeren HR, Deuter CE, Joerissen JD, Schroder A, Otte C, Wingenfeld K. Decision making in response to physiological and combined physiological and psychosocial stress. Behav Neurosci. 2019 Feb;133(1):59-67. doi: 10.1037/bne0000288. Epub 2018 Dec 17. PMID 30556701
- [Background] Wilson MH, Newman S, Imray CH. The cerebral effects of ascent to high altitudes. Lancet Neurol. 2009 Feb;8(2):175-91. doi: 10.1016/S1474-4422(09)70014-6. PMID 19161909
- [Derived] Falla M, van Veelen MJ, Falk M, Weiss EM, Roveri G, Mase M, Weber B, Randi A, Brugger H, Hufner K, Strapazzon G. Effect of oxygen supplementation on cognitive performance among HEMS providers after acute exposure to altitude: the HEMS II randomized clinical trial. Scand J Trauma Resusc Emerg Med. 2024 Jul 29;32(1):65. doi: 10.1186/s13049-024-01238-6. PMID 39075543